CLINICAL TRIAL: NCT06561971
Title: Evaluating the Effect of Smoking Amount on Determining Salivary High Sensitive C-Reactive Protein(Hs-CRP) Values by Centrifuging the Saliva of the Same Individuals at Different Rpm and Time.
Brief Title: Effect of Different Centrifuge Values on Saliva High Sensitive C-Reactive Protein (Hs-CRP) Levels in Individuals With Different Smoking Amounts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ece Ozer, Research Assistant, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-SAEK-0029
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: According to full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL),bleeding on probing (BOP), gingival index (GI) and plaque index (PI) samples of saliva were obtained from 90 systemically healthy non-smoker individuals with heavy smokers (H, n=30), light smokers(L, n=30) and non-smokers (N, n=30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-Smokers (Experimental): Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: saliva obtaining
- Light Smokers (Experimental): Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: saliva obtaining
- Heavy Smokers (Experimental): Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: saliva obtaining

INTERVENTIONS:
Diagnostic Test: saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated saliva was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Tubes were stored at -80ºC until the day of analysis.

SUMMARY:
The purpose of this study; In periodontally healthy individuals, high sensitive c-reactive protein (hs-CRP) levels of non-smokers, smokers of less than 10 cigarettes per day and smokers of more than 10 cigarettes per day were measured at 15 rpm-10 min, 10 centrifuge values, which are frequently used in saliva studies. To determine the levels in saliva samples as a result of rpm-10 min and 10 rpm 6 min centrifugations and to determine the values at which a cytokine of this molecular weight should be centrifuged and to examine the possible correlation between these values and the clinical parameters of the amount of smoking. Materials and Methods: saliva samples were collected from 90 systemically healthy individuals who were non-smokers (N, n=30), light smokers <10 cigarettes per day (L, n=30) and heavy smokers >10 cigarettes per day (H, n=20). samples were taken. Full-mouth clinical periodontal measurements, including probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP), gingival index (GI), and plaque index (PI), were also recorded. Enzyme-linked immunosorbent assay (ELISA) was used to determine hs-CRP levels in biological samples.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Periodontally clinical healthy
* At least 20 permanent teeth in the mouth
* No medication for continuous use
* Those who have not used antibiotics, anti-inflammatory and systemic corticosteroid drugs in the last 6 months.
* Not in pregnancy or lactation period.
* Not received periodontal treatment in the last 6 months

  * For the non-smoker group; person who does not smoke tobacco
  * For the light-smoker group; person who smokes less than 10 cigarettes a day
  * For heavy-smoker group; person who smokes more than 10 cigarettes a day

Exclusion Criteria:

* Any oral or systemic disease
* Regularly using a systemic medication
* During pregnancy or lactation
* Received periodontal treatment within the last 6 months.
* Those who received antibiotic, anti-inflammatory or systemic corticosteroid medication in the last 6 months
* Individual with periodontal disease

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-01-22 (Estimated)

PRIMARY OUTCOMES:
The total amount of hs-CRP in saliva | 24 hours after taking the clinical measurements at the first visit

SECONDARY OUTCOMES:
Determining the ideal centrifugal value range of hs-CRP saliva level | Within 1 week after receiving the biochemical analysis results

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Çelebi University Department of Periodontology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol